CLINICAL TRIAL: NCT00498927
Title: A Phase II Trial of Continuous Low-Dose Temozolomide for Patients With Recurrent Malignant Glioma
Brief Title: Temozolomide in Treating Patients With Recurrent Glioblastoma Multiforme or Other Malignant Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Weill Medical College of Cornell University (Other); Schering-Plough (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-064; P30CA008748 (NIH); MSKCC-07064; SPRI-PO5096
Record Dates: First submitted 2007-07-10; First posted 2007-07-11 (Estimated); Results first posted 2016-02-29 (Estimated); Last update posted 2016-02-29 (Estimated); Status verified 2016-02

CONDITIONS: Brain and Central Nervous System Tumors
Keywords: recurrent adult brain tumor; adult giant cell glioblastoma; adult glioblastoma; adult gliosarcoma; adult anaplastic astrocytoma; adult diffuse astrocytoma; adult pilocytic astrocytoma; adult subependymal giant cell astrocytoma; adult anaplastic ependymoma; adult ependymoma; adult myxopapillary ependymoma; adult subependymoma; adult anaplastic oligodendroglioma; adult oligodendroglioma; adult brain stem glioma; adult mixed glioma; adult pineal gland astrocytoma
MeSH Terms: conditions — Central Nervous System Neoplasms; Brain Neoplasms; Glioblastoma; Gliosarcoma; Astrocytoma; Ependymoma; Glioma, Subependymal; Oligodendroglioma; Glioma | interventions — Temozolomide; Reverse Transcriptase Polymerase Chain Reaction; Immunoenzyme Techniques

ARMS (1):
- Temozolomide (Experimental): Following diagnosis of tumor recurrence or progression, all patients will receive of daily low dose temozolomide given at 50mg/m2/d without interruption. Brain imaging will be performed at baseline and every 2 months (standard of care). The treatment will be administered until development of toxicity, evidence of progression of disease or death.
  Interventions: Drug: temozolomide; Genetic: protein expression analysis; Genetic: reverse transcriptase-polymerase chain reaction; Other: diagnostic laboratory biomarker analysis; Other: immunoenzyme technique

INTERVENTIONS:
Drug: temozolomide
Genetic: protein expression analysis
Genetic: reverse transcriptase-polymerase chain reaction
Other: diagnostic laboratory biomarker analysis
Other: immunoenzyme technique

SUMMARY:
RATIONALE: Drugs used in chemotherapy, such as temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing.

PURPOSE: This phase II trial is studying how well temozolomide works in treating patients with recurrent glioblastoma multiforme or other malignant glioma.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the progression-free survival rate at 6 months in patients with recurrent glioblastoma multiforme or other malignant glioma treated with temozolomide.

Secondary

* Determine the overall survival of patients treated with this drug.

OUTLINE: Patients receive oral temozolomide once daily in the absence of disease progression or unacceptable toxicity.

Blood samples are collected at baseline and every 2 months for 2 years for evaluation of markers of neo-angiogenesis. Samples are analyzed by protein expression, reverse-transcriptase PCR, ELISA, and western blot. (Samples are no longer being collected and tested as of 1/12/09)

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Pathologically diagnosed glioblastoma multiforme or other malignant glioma

  * Recurrent disease
* Must have received prior temozolomide

PATIENT CHARACTERISTICS:

* Karnofsky performance status 60-100%
* Granulocyte count ≥ 1,500/mm³
* Platelet count ≥ 100,000/mm³
* SGOT ≤ 2.5 times upper limit of normal (ULN)
* Creatinine ≤ 2 times ULN
* Bilirubin ≤ 2 times ULN
* No other active malignancy except for cervical carcinoma in situ or basal cell carcinoma of the skin
* No serious medical or psychiatric illness that, in the opinion of the investigator, would preclude study treatment
* No medical condition that precludes swallowing pills
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* Recovered from all prior therapy

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2007-06; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Antonio Omuro, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center; Thomas Kaley, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

REFERENCES:
- [Derived] Omuro A, Chan TA, Abrey LE, Khasraw M, Reiner AS, Kaley TJ, Deangelis LM, Lassman AB, Nolan CP, Gavrilovic IT, Hormigo A, Salvant C, Heguy A, Kaufman A, Huse JT, Panageas KS, Hottinger AF, Mellinghoff I. Phase II trial of continuous low-dose temozolomide for patients with recurrent malignant glioma. Neuro Oncol. 2013 Feb;15(2):242-50. doi: 10.1093/neuonc/nos295. Epub 2012 Dec 14. PMID 23243055

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Temozolomide
Started | 47
Completed | 47
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Temozolomide
Number analyzed (Participants) | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 36
  >=65 years | 11
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 31

OUTCOME MEASURES:

1. Primary Outcome: Progression-free Survival (PFS) Rate at 6 Months
Description: Progression is defined using Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0), as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions.
Time Frame: at 6 months
Population: Glioblastoma patients
Measure: Number; unit: percentage of participants
Arm/Group | Temozolomide
Number analyzed (Participants) | 37
percentage of participants | 19

2. Secondary Outcome: Overall Survival
Description: All patients will have their tumor measurements recorded at baseline and at the time of each MRI scan. Lesions must be measured in two dimensions. The dose of gadolinium must be held constant from scan to scan. Macdonald criteria will be used for assessment of tumor response.
Time Frame: 2 years
Population: Glioblastoma patients
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Temozolomide
Number analyzed (Participants) | 37
months | 7 [5 to 12]

ADVERSE EVENTS:
Arm/Group | Temozolomide
Serious Adverse Events (participants affected / at risk) | 14/47
Other Adverse Events (participants affected / at risk) | 14/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide (N=47)
AST, SGOT (Blood and lymphatic system disorders) | 1 (1)
CNS cerebrovascular ischemia (Nervous system disorders) | 1 (1)
Cognitive disturbance (Nervous system disorders) | 1 (1)
Confusion (General disorders) | 3 (3)
Extremity-lower (gait/walking) (General disorders) | 2 (2)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 2 (2)
Infection, other (Infections and infestations) | 1 (1)
Mood alteration - Agitation (General disorders) | 1 (1)
Pain - Back (General disorders) | 1 (1)
Pain - Head/headache (General disorders) | 2 (2)
Pyramidal tract dysfunction (Nervous system disorders) | 1 (1)
Seizure (General disorders) | 2 (2)
Speech impairment (General disorders) | 1 (1)
Thrombosis/thrombus/embolism (Cardiac disorders) | 1 (1)
Dehydration (Gastrointestinal disorders) | 1 (1)
Neurology - Other (specify) (Nervous system disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Temozolomide (N=47)
Fatigue (asthenia, lethargy, malaise) (General disorders) | 3 (3)
Glucose, high (hyperglycemia) (Metabolism and nutrition disorders) | 7 (7)
Leukocytes (total WBC) (Blood and lymphatic system disorders) | 6 (6)
Lymphopenia (Blood and lymphatic system disorders) | 7 (7)
Neuropathy: sensory (Nervous system disorders) | 3 (3)
Platelets (Blood and lymphatic system disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes